CLINICAL TRIAL: NCT04876833
Title: Characteristics of Intestinal Microbiome in the Progression of Early Chronic Obstructive Pulmonary Disease
Brief Title: Characteristics of Intestinal Microbiome in the Progression of Early COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: MR-61-21-012951
Record Dates: First submitted 2021-04-25; First posted 2021-05-07 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Intestinal Microbiome; Metabolite; Immune Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Fecal Specimen,Serum Specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HC，healthy control: 18-65 years old，no smoking history，normal pulmonary function，normal compatible computed tomography.
- HG，high-risk COPD group: 18-60 years old，≥10 pack-years smoking history，normal pulmonary function，normal compatible computed tomography.
- EG，early COPD group: 18-60 years old，≥10 pack-years smoking history，and with any of the following abnormalities：
  1. Forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) less than 80%;
  2. Compatible computed tomography abnormalities：airway abnormality and/or emphysema，air trapping, or bronchial thickening；
  3. FEV1 decline (≥60 mL per year).
- MG，mild and moderate COPD group: 18-65 years old，FEV1/FVC<70%，FEV1%predicted ≥50%.

SUMMARY:
This study is aiming at explore the characteristics of intestinal microbiome during the early progression of COPD, the correlation between the changes of intestinal microbiome and the severity and risk of acute exacerbation of COPD, the correlation between microbial metabolites SCFA and immune function of COPD. Then reveal the influence of intestinal microecology on the development of COPD and the possible mechanism of intestinal microecology in the pathogenesis of COPD.

DETAILED DESCRIPTION:
1. Invite participants according to inclusion criteria and exclusion criteria and divide them into 4 groups, including healthy control (HC), high-risk COPD group (HG), early COPD group (EG), mild and moderate COPD group (MG). Research contents will be explained detailedly to the participants, and the healthy participants and COPD patients who volunteer to participate in this study will sign the informed consent form (ICF) under the premise of adequate understanding.
2. Collect clinical data of the participants and asses the severity of symptoms and the risk of acute exacerbation of COPD patients. Clinical data include general condition, history of past illness, history of present illness, personal history, family history and the examination results of blood routine, pulmonary function and compatible computed tomography. Breathlessness measurement adopt the modified British Medical Reseach Council (mMRC); symptoms measurement adopt COPD assessment test (CAT); quality of life measurement adopt St. George's Respiratory Questionnaire (SGRQ); risk of acute exacerbation measurement adopt dyspnea，degree of airflow obstruction，smoking status and the number of exacerbation (DOSE) scoring system.
3. Collect fecal specimens from the participants on the morning of the same day. During the first three days of collection, they should keep their daily dietary habits and avoid sudden changes in dietary habits. Considerations: first remove the urine, excrement into a clean dry container, do not mix with urine and other sundries; the part of the feces that do not contact the air and container is taken from the specimen; women who are menstruating cannot be sampled. Each participant collect 3 fecal samples with a sterile spoon in a sterile enzyme-free cryopreservation tube, label the sample name and date, quickly placed in a -20℃ refrigerator, and transported to the hospital within 2 hours, where they were stored at -80℃. Fecal microbiome are detected by 16S rRNA gene sequencing and metabolite short chain fatty acid (SCFA) are detected by Gaschromatography (GC).
4. Serum of participants are collected at the clinical laboratory and detect indicators related to immune function by enzyme-linked immunosorbent assay (ELISA).
5. Explore the characteristics of intestinal microbiome during the early progression of COPD, the correlation between the changes of intestinal microbiome and the severity and risk of acute exacerbation of COPD, the correlation between microbial metabolites SCFA and immune function of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. ≥10 pack-years smoking history;
2. Examination of pulmonary function and compatible computed tomography meeting group requirements (as shown in Groups and Interventions).

Exclusion Criteria:

1. Take antibiotics, probiotics, prebiotics, synbiotics and other drugs that obviously interfere with intestinal microbiome within 2 months;
2. Suffer from other chronic respiratory diseases other than COPD (such as bronchial asthma, allergic rhinitis, pulmonary interstitial fibrosis, bronchiectasis, lung cancer, etc.);
3. Suffer from severe intestinal diseases (such as inflammatory bowel disease, intestinal infections, colorectal cancer, etc.);
4. Suffer from serious hematopoietic system diseases, and the brain, heart, liver, kidney and other important organs are damaged;
5. Suffer from severe hypertension, coronary heart disease, diabetes and other chronic diseases and taking drugs for long-term maintenance;
6. Suffer from active infectious diseases (hepatitis B, tuberculosis, etc.);
7. Pregnant or lactating women;
8. Patients with obvious anxiety, depression and other psychiatric symptoms and patients with schizophrenia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are from Physical Examination Department and Respiratory and Critical Care Medicine Department of the Second Affiliated Hospital of Xi 'an Jiaotong University.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Breathlessness measurement | 1 month
  modified British Medical Reseach Council (mMRC)：the score increases from 0 to 4，and higher scores mean a heavier symptom.
Symptoms measurement | 1 month
  COPD assessment test (CAT)：the score increases from 0 to 40，and higher scores mean a heavier symptom.
Quality of life measurement | 1 month
  St. George's Respiratory Questionnaire (SGRQ): the score increases from 0 to 100，and higher scores mean a heavier symptom.
Risk of acute exacerbation of participants | 1 month
  dyspnea，degree of airflow obstruction，smoking status，the number of exacerbation (DOSE): the score increases from 0 to 9，and higher scores mean a higher risk of acute exacerbation.
Pulmonary function | 1 month
  Forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC), FEV1%predicted, MMEF25-75%: range from 0%-100%, and higher percentages mean a heavier symptom.
Compatible computed tomography | 1 month
  mean lung density
Characteristics of intestinal microbiome | 1 month
  Alpha diversity，Beta diversity，Species differences between groups at different taxonomic levels.
Contents of short chain fatty acid in fecal samples | 1 month
  acetic acid, propionic acid, butyric acid
Blood routine | 1 month
  neutrophilic granulocyte percent, eosinophilic granulocyte percent: higher percentages mean a heavier symptom.
Concentration of protein in serum | 1 month
  fibrinogen, C-reactive protein, surfactant protein-D(SP-D)
Concentration of enzyme in serum | 1 month
  neutrophil elastase, alpha1-antitrypsin
Concentration of inflammatory factor in serum | 1 month
  TNF-α, IFN-γ, IL-6, IL-8, IL-17
Concentration of chemokine in serum | 1 month
  CCL-16, CCL-18

CONTACTS AND LOCATIONS:
Overall Officials: Yun Liu, MD, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share with others the deidentified individual-patient data (IPD) underlying the results presented in the article (including tables, figures, and appendices or supplementary material).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication; no end date
Access Criteria: We plan to share with anyone who wishes to access the data for any purpose of analyses and data are available indefinitely.

REFERENCES:
- [Background] Tsay JJ, Segal LN. Could the Sputum Microbiota Be a Biomarker That Predicts Mortality after Acute Exacerbations of Chronic Obstructive Pulmonary Disease? Am J Respir Crit Care Med. 2019 May 15;199(10):1175-1176. doi: 10.1164/rccm.201811-2138ED. No abstract available. PMID 30485116
- [Background] Stockley RA, Halpin DMG, Celli BR, Singh D. Chronic Obstructive Pulmonary Disease Biomarkers and Their Interpretation. Am J Respir Crit Care Med. 2019 May 15;199(10):1195-1204. doi: 10.1164/rccm.201810-1860SO. PMID 30592902
- [Background] Budden KF, Gellatly SL, Wood DL, Cooper MA, Morrison M, Hugenholtz P, Hansbro PM. Emerging pathogenic links between microbiota and the gut-lung axis. Nat Rev Microbiol. 2017 Jan;15(1):55-63. doi: 10.1038/nrmicro.2016.142. Epub 2016 Oct 3. PMID 27694885
- [Result] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Result] Wang C, Xu J, Yang L, Xu Y, Zhang X, Bai C, Kang J, Ran P, Shen H, Wen F, Huang K, Yao W, Sun T, Shan G, Yang T, Lin Y, Wu S, Zhu J, Wang R, Shi Z, Zhao J, Ye X, Song Y, Wang Q, Zhou Y, Ding L, Yang T, Chen Y, Guo Y, Xiao F, Lu Y, Peng X, Zhang B, Xiao D, Chen CS, Wang Z, Zhang H, Bu X, Zhang X, An L, Zhang S, Cao Z, Zhan Q, Yang Y, Cao B, Dai H, Liang L, He J; China Pulmonary Health Study Group. Prevalence and risk factors of chronic obstructive pulmonary disease in China (the China Pulmonary Health [CPH] study): a national cross-sectional study. Lancet. 2018 Apr 28;391(10131):1706-1717. doi: 10.1016/S0140-6736(18)30841-9. Epub 2018 Apr 9. PMID 29650248
- [Result] Colak Y, Afzal S, Nordestgaard BG, Vestbo J, Lange P. Prevalence, Characteristics, and Prognosis of Early Chronic Obstructive Pulmonary Disease. The Copenhagen General Population Study. Am J Respir Crit Care Med. 2020 Mar 15;201(6):671-680. doi: 10.1164/rccm.201908-1644OC. PMID 31770495
- [Result] Bowerman KL, Rehman SF, Vaughan A, Lachner N, Budden KF, Kim RY, Wood DLA, Gellatly SL, Shukla SD, Wood LG, Yang IA, Wark PA, Hugenholtz P, Hansbro PM. Disease-associated gut microbiome and metabolome changes in patients with chronic obstructive pulmonary disease. Nat Commun. 2020 Nov 18;11(1):5886. doi: 10.1038/s41467-020-19701-0. PMID 33208745
- [Result] Jang YO, Lee SH, Choi JJ, Kim DH, Choi JM, Kang MJ, Oh YM, Park YJ, Shin Y, Lee SW. Fecal microbial transplantation and a high fiber diet attenuates emphysema development by suppressing inflammation and apoptosis. Exp Mol Med. 2020 Jul;52(7):1128-1139. doi: 10.1038/s12276-020-0469-y. Epub 2020 Jul 17. PMID 32681029
- [Result] Sprooten RTM, Lenaerts K, Braeken DCW, Grimbergen I, Rutten EP, Wouters EFM, Rohde GGU. Increased Small Intestinal Permeability during Severe Acute Exacerbations of COPD. Respiration. 2018;95(5):334-342. doi: 10.1159/000485935. Epub 2018 Jan 25. PMID 29393240
- [Result] Keely S, Talley NJ, Hansbro PM. Pulmonary-intestinal cross-talk in mucosal inflammatory disease. Mucosal Immunol. 2012 Jan;5(1):7-18. doi: 10.1038/mi.2011.55. Epub 2011 Nov 16. PMID 22089028
- [Result] Wypych TP, Wickramasinghe LC, Marsland BJ. The influence of the microbiome on respiratory health. Nat Immunol. 2019 Oct;20(10):1279-1290. doi: 10.1038/s41590-019-0451-9. Epub 2019 Sep 9. PMID 31501577
- [Result] Mortaz E, Adcock IM, Ricciardolo FL, Varahram M, Jamaati H, Velayati AA, Folkerts G, Garssen J. Anti-Inflammatory Effects of Lactobacillus Rahmnosus and Bifidobacterium Breve on Cigarette Smoke Activated Human Macrophages. PLoS One. 2015 Aug 28;10(8):e0136455. doi: 10.1371/journal.pone.0136455. eCollection 2015. PMID 26317628
- [Result] Reale M, Boscolo P, Bellante V, Tarantelli C, Di Nicola M, Forcella L, Li Q, Morimoto K, Muraro R. Daily intake of Lactobacillus casei Shirota increases natural killer cell activity in smokers. Br J Nutr. 2012 Jul;108(2):308-14. doi: 10.1017/S0007114511005630. Epub 2011 Dec 6. PMID 22142891
- [Result] Tomoda K, Kubo K, Dairiki K, Yamaji T, Yamamoto Y, Nishii Y, Nakamura A, Yoshikawa M, Hamada K, Kimura H. Whey peptide-based enteral diet attenuated elastase-induced emphysema with increase in short chain fatty acids in mice. BMC Pulm Med. 2015 Jun 10;15:64. doi: 10.1186/s12890-015-0059-2. PMID 26059026
- [Result] Lee SH, Yun Y, Kim SJ, Lee EJ, Chang Y, Ryu S, Shin H, Kim HL, Kim HN, Lee JH. Association between Cigarette Smoking Status and Composition of Gut Microbiota: Population-Based Cross-Sectional Study. J Clin Med. 2018 Sep 14;7(9):282. doi: 10.3390/jcm7090282. PMID 30223529
- [Result] Li N, Yang Z, Liao B, Pan T, Pu J, Hao B, Fu Z, Cao W, Zhou Y, He F, Li B, Ran P. Chronic exposure to ambient particulate matter induces gut microbial dysbiosis in a rat COPD model. Respir Res. 2020 Oct 19;21(1):271. doi: 10.1186/s12931-020-01529-3. PMID 33076910
- See also: Correlation index analysis of intestinal flora and inflammatory factors in patients with chronic obstructive pulmonary disease — https://d.wanfangdata.com.cn/periodical/ChlQZXJpb2RpY2FsQ0hJTmV3UzIwMjEwNDE1EhFsaW5janl6ejIwMjAwMTAzNhoIbzR0Y24zenE%3D
- See also: Characteristics of intestinal flora in patients with chronic obstructive pulmonary disease and their correlation with inflammatory markers and pulmonary function status — https://d.wanfangdata.com.cn/periodical/ChlQZXJpb2RpY2FsQ0hJTmV3UzIwMjEwNDE1EhFsaW5janl6ejIwMjAwMTAzNhoIajdrcWM1dXA%3D